CLINICAL TRIAL: NCT00110305
Title: A Phase IIb Randomized, Partially Blinded, Dose-Finding Trial of TMC278 in Antiretroviral-Naive HIV-1 Infected Subjects
Brief Title: A Study of TMC278 in Human Immunodeficiency Virus Type 1 Infected Patients, Who Are Not Treated With Antiretroviral Medicines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006760; TMC278-C204 (Other: Tibotec Pharmaceuticals, Ireland); R278474-C204 (Other: Tibotec Pharmaceuticals, Ireland); NCT00980837 (obsolete NCT alias)
Record Dates: First submitted 2005-05-05; First posted 2005-05-06 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Human Immunodeficiency Virus Type 1; Human immunodeficiency virus (HIV); Antiretroviral; Antiviral; ARV; TMC278; Efavirenz; Combivir; Truvada; Zidovudine; Lamivudine; Tenofovir disoproxil fumarate; Emtricitabine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Rilpivirine; efavirenz; lamivudine, zidovudine drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TMC278 25 mg (Experimental): Participants will receive TMC278 25 mg once daily up to Week 96. Later on, participants will receive TMC278 75 mg once daily up to Week 144 and then TMC278 25 mg once daily up to Week 240.
  Interventions: Drug: TMC278 25 mg; Drug: Non-nucleoside reverse transcriptase inhibitor (NRTIs)
- TMC278 75 mg (Experimental): Participants will receive TMC278 75 mg once daily up to Week 144. Later on, participants will receive TMC278 25 mg once daily up to Week 240.
  Interventions: Drug: TMC278 75 mg; Drug: Non-nucleoside reverse transcriptase inhibitor (NRTIs)
- TMC278 150 mg (Experimental): Participants will receive TMC278 150 mg once daily up to Week 96. Later on, participants will receive TMC278 75 mg once daily up to Week 144 and then TMC278 25 mg once daily up to Week 240.
  Interventions: Drug: TMC278 150 mg; Drug: Non-nucleoside reverse transcriptase inhibitor (NRTIs)
- Efavirenz (Active Comparator): Participants will receive efavirenz 600 mg once daily up to Week 96. Later on, participants will have an option to continue on efavirenz until Week 144 or until Week 240.
  Interventions: Drug: Efavirenz; Drug: Non-nucleoside reverse transcriptase inhibitor (NRTIs)

INTERVENTIONS:
Drug: TMC278 25 mg — TMC278 25 mg tablet will be administered once daily.
  Arms: TMC278 25 mg
Drug: TMC278 75 mg — TMC278 75 mg (1 X 25 mg + 1 X 50 mg) tablets will be administered once daily.
  Arms: TMC278 75 mg
Drug: TMC278 150 mg — TMC278 150 mg (1 X 50 mg + 1 X 100 mg) tablets will be administered once daily.
  Arms: TMC278 150 mg
Drug: Efavirenz — Efavirenz 600 mg (1 x 600 mg tablet or 3 x 200 mg capsules, depending on formulation locally available) will be administered once daily.
  Arms: Efavirenz
Drug: Non-nucleoside reverse transcriptase inhibitor (NRTIs) — Investigator selected 2 NRTIs: (1) Zidovudine and lamivudine (Combivir) and (2) tenofovir disoproxil fumarate and emtricitabine (Truvada) will be administered as per the package inserts, along with the TMC278 during the study period.
  Other Names: Combivir; Truvada

SUMMARY:
The purpose of this study is to evaluate the dose-response relationship of antiviral activity after 48 weeks treatment with 3 different dose regimens of TMC278.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), active controlled (participants are assigned to either a recognized effective treatment or the study medication) study. This study consists of 3 phases: screening phase (4 weeks), treatment phase (96 weeks), and follow up phase (4 weeks). In the treatment phase, participants will be randomly assigned to 1 of the 4 treatment groups: (1) TMC278 25 mg, (2) TMC278 75 mg, (3) TMC278 150 mg, or (4) efavirnez (control group); along with investigator selected 2 non-nucleoside reverse transcriptase inhibitor (NRTIs) until Week 96. TMC278 will be assigned by double-blinded fashion (participant and investigator are not aware of the TMC278 dose what participants will receive) and efavirnez will be assigned by open-label fashion (all people know what treatment participants will receive). After Week 96, 3 optional open-label (all people know the identity of the intervention) extension periods will be conducted to collect long term safety and effectiveness data of TMC278. 3 optional extension periods are: first optional extension period (all participants will receive TMC278 75 mg + 2 NRTIs from Week 96 to Week144); second optional extension period (all participants will receive TMC278 25 mg + 2 NRTIs from Week 144 to Week 240); and third optional extension period (all participants will receive TMC278 25 mg + 2 NRTIs from Week 240 until TMC278 is commercially available). Participants on efavirenz group will have the option to continue on efavirenz + 2 NRTIs until the total treatment duration of 240 weeks. Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, physical examination, and vital signs which will be monitored throughout the study. The maximum duration of the study will be 104, 152, or 248 weeks, plus the optional third extension period.

ELIGIBILITY:
Inclusion Criteria:

* Documented human immunodeficiency virus type 1 (HIV-1) infection
* Never been treated with an antiretroviral (ARV) treatment or therapeutic HIV vaccine, or received less than or equal to 2 weeks treatment prior to screening with an nucleoside reverse transcriptase inhibitors
* HIV-1 plasma viral load above 5000 HIV-1 RNA copies per milliliter, at screening
* Cortisol of at least 550 nano moles per liter (19.9 microgram per deciliter) at screening
* Sensitivity to investigator selected nucleosides, at screening

Exclusion Criteria:

* Currently having active Acquired Immunodeficiency Syndrome (AIDS) defining illness
* Known or suspected acute (primary) HIV-1 infection
* Any current or history of adrenal disorder, and an acute hepatitis A, B, or C infection
* Documented genotypic evidence of Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) resistance at screening
* Pregnant or breastfeeding females
* Not agree to protocol-defined effective use of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2005-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (40):
- United States (9):
  - Beverly Hills, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Addison, Texas
  - Seattle, Washington
- Argentina (2):
  - Buenos Aires
  - Rosario
- Vienna, Austria
- Brazil (5):
  - Campinas
  - Curitiba
  - Pinheiros
  - Rio de Janeiro
  - São Paulo
- Beijing, China
- France (2):
  - Paris
  - Tourcoing
- Germany (4):
  - Berlin
  - Cologne
  - Freiburg im Breisgau
  - München
- Mexico City, Mexico
- San Juan, Puerto Rico
- Russia (5):
  - Kazan'
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Volgograd
- South Africa (3):
  - Bloemfontein
  - Cape Town
  - Johannesburg
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Kampala, Uganda
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- [Derived] Pozniak AL, Morales-Ramirez J, Katabira E, Steyn D, Lupo SH, Santoscoy M, Grinsztejn B, Ruxrungtham K, Rimsky LT, Vanveggel S, Boven K; TMC278-C204 Study Group. Efficacy and safety of TMC278 in antiretroviral-naive HIV-1 patients: week 96 results of a phase IIb randomized trial. AIDS. 2010 Jan 2;24(1):55-65. doi: 10.1097/QAD.0b013e32833032ed. PMID 19926964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 368 participants were enrolled at multiple centers in different countries.
Pre-assignment Details: 368 participants were randomly assigned to 4 treatment groups (TMC278 25 mg: 93; TMC278 75 mg: 95; TMC278 150 mg: 91; and Efavirenz: 89). Participant flow through Week 240 was reported for the combined TMC278 and Efavirenz groups, as all TMC278 participants were switched after Week 96 initially to 75 mg and subsequently to 25 mg dose.
Groups:
- All TMC278: TMC278 25 mg, 75 mg, and 150 mg once daily
- Efavirenz: Efavirenz 600 mg once daily
Period: Overall Study
Arm/Group | All TMC278 | Efavirenz
Started | 279 | 89
Completed | 165 | 57
Not Completed | 114 | 32
Not completed — Adverse Event | 46 | 13
Not completed — Sponsors Decision | 1 | 0
Not completed — Subject Non-Compliant | 9 | 2
Not completed — Subject Ineligible To Continue The Trial | 2 | 1
Not completed — Subject Reached A Virologic Endpoint | 21 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 20 | 3
Not completed — Other | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- TMC278 25 mg: TMC278 25 mg once daily
- TMC278 75 mg: TMC278 75 mg once daily
- TMC 150 mg: TMC278 150 mg once daily
- Total: Total of all reporting groups
Arm/Group | TMC278 25 mg | TMC278 75 mg | TMC 150 mg | Efavirenz | Total
Number analyzed (Participants) | 93 | 95 | 91 | 89 | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 92 | 95 | 89 | 89 | 365
  >=65 years | 1 | 0 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.9) | 36.3 (8.3) | 35.9 (9.7) | 35.4 (8.1) | 36.1 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 33 | 29 | 121
  Male | 65 | 64 | 58 | 60 | 247
Region Enroll [Number; unit: participants]
  Asia, South Africa and Uganda | 32 | 32 | 31 | 29 | 124
  Europe, USA and Russia | 33 | 33 | 32 | 32 | 130
  Latin America | 28 | 30 | 28 | 28 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Response at Week 48 (Viral Load Less Than 50 Copies Per mL) - as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: The TLOVR algorithm was used to derive response, ie, response and loss of response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders. Participants with intermittent missing viral load values were considered responders if the preceeding and succeeding visits indicated response. In all other cases, intermittent values were imputed with nonresponse. Resuppression after confirmed virologic failure was considered as failure in this algorithm.
Time Frame: Week 48
Population: Intent to treat population: Participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Groups:
- TMC278 150 mg: TMC278 150 mg once daily
- Efavirenz: Efaviren 600 mg once daily
Arm/Group | TMC278 25 mg | TMC278 75 mg | TMC278 150 mg | All TMC278 | Efavirenz
Number analyzed (Participants) | 93 | 95 | 91 | 279 | 89
Participants | 74 | 76 | 70 | 220 | 72
Statistical Analysis 1: Comparison: TMC278 25 mg vs TMC278 75 mg; Test type: Superiority or Other; p = 0.92, Regression, Logistic — The significance level for each comparison was 5% (two-sided). No further adjustment of this significance level was applied; This model with factors treatment, region, and Nucleoside/tide reverse transcriptase inhibitors (N[t]RTIs) used, and baseline viral load as covariate; Differences in response rate = 0.5, 95% CI 2-sided [-10.4 to 11.3]
Statistical Analysis 2: Comparison: TMC278 25 mg vs TMC278 150 mg; Test type: Superiority or Other; p = 0.56, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; This model with factors treatment, region, and N(t)RTIs used, and baseline viral load as covariate; Difference in response rate = -2.3, 95% CI 2-sided [-13.6 to 9.0]
Statistical Analysis 3: Comparison: TMC278 75 mg vs TMC278 150 mg; Test type: Superiority or Other; p = 0.62, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; This model with factors treatment, region, and N(t)RTIs used, and baseline viral load as covariate; Difference in response rate = -2.8, 95% CI 2-sided [-14.0 to 8.4]
Statistical Analysis 4: Comparison: All TMC278 vs Efavirenz; Test type: Superiority or Other; p = 0.80, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; This model with factors treatment, region, and N(t)RTIs used, and baseline viral load as covariate; Difference in response rate = -1.5, 95% CI 2-sided [-10.5 to 7.5]

2. Secondary Outcome: Number of Participants With Virologic Response at Week 96 (Viral Load Less Than 50 Copies Per mL) - as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: as for outcome 1
Time Frame: Week 96
Population: Intent to treat population: Participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | TMC278 25 mg | TMC278 75 mg | TMC278 150 mg | All TMC278 | Efavirenz
Number analyzed (Participants) | 93 | 95 | 91 | 279 | 89
Participants | 71 | 68 | 65 | 204 | 63
Statistical Analysis 1: Comparison: TMC278 25 mg vs TMC278 75 mg; Test type: Superiority or Other; p = 0.45, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in response rate = -4.8, 95% CI 2-sided [-17.1 to 7.6]
Statistical Analysis 2: Comparison: TMC278 25 mg vs TMC278 150 mg; Test type: Superiority or Other; p = 0.45, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; This model with factors treatment, region, and N(t)RTIs used, and baseline viral load as covariate; Difference in response rate = -4.8, 95% CI 2-sided [-17.3 to 7.7]
Statistical Analysis 3: Comparison: TMC278 75 mg vs TMC278 150 mg; Test type: Superiority or Other; p = 0.99, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; This model with factors treatment, region, and N(t)RTIs used, and baseline viral load as covariate; Difference in response rate = 0.0, 95% CI 2-sided [-12.9 to 12.8]
Statistical Analysis 4: Comparison: All TMC278 vs Efavirenz; Test type: Superiority or Other; p = 0.63, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; This model with factors treatment, region, and N(t)RTIs used, and baseline viral load as covariate; Differences in response = 2.6, 95% CI 2-sided [-8.1 to 13.3]

3. Secondary Outcome: Number of Participants With Virologic Response at Week 96 (Viral Load Less Than 50 Copies Per mL) - Snapshot Analysis
Description: The analysis is based on the last observed viral load data within the Week 96 window. Virologic response is defined as a viral load less than 50 copies/mL. Missing viral load was considered as non-response.
Time Frame: Week 96
Population: Intent to treat population: Participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | TMC278 25 mg | TMC278 75 mg | TMC278 150 mg | All TMC278 | Efavirenz
Number analyzed (Participants) | 93 | 95 | 91 | 279 | 89
Participants | 71 | 70 | 66 | 207 | 64

4. Secondary Outcome: Number of Participants With Virologic Response at Week 240 (Viral Load Less Than 50 Copies Per mL) - as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: as for outcome 1
Time Frame: Week 240
Population: Intent to treat population: Participants who received at least 1 dose of study medication. This was measured at Week 240 for the combined TMC278 and Efavirenz groups, as all TMC278 participants were switched after Week 96 initially to 75 mg and subsequently to 25 mg dose.
Measure: Number; unit: Participants
Arm/Group | All TMC278 | Efavirenz
Number analyzed (Participants) | 279 | 89
Participants | 152 | 51
Statistical Analysis 1: Comparison: All TMC278 vs Efavirenz; Test type: Superiority or Other; Difference in response rate = -2.8, 95% CI [-14.7 to 9.1]

5. Secondary Outcome: Number of Participants With Virologic Response at Week 240 (Viral Load Less Than 50 Copies Per mL) - Snapshot Analysis
Description: The analysis is based on the last observed viral load data within the Week 240 window. Virologic response is defined as a viral load less than 50 copies/mL. Missing viral load was considered as non-response.
Time Frame: Week 240
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | All TMC278 | Efavirenz
Number analyzed (Participants) | 279 | 89
Participants | 150 | 51

6. Secondary Outcome: Number of Participants With Virologic Response at Week 240 (Viral Load Less Than 400 Copies/mL) - as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: as for outcome 1
Time Frame: Week 240
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | All TMC278 | Efavirenz
Number analyzed (Participants) | 279 | 89
Participants | 166 | 54

7. Secondary Outcome: Change From Baseline in CD4+ Cell Count (Absolute) at Week 96
Description: Change from baseline in CD4+ cell count was imputed in case of missing values: in case of premature discontinuation, data were imputed with the baseline value after discontinuation (i.e. change=0, Non-Completer [NC] = Failure); otherwise last observation carried forward was applied.
Time Frame: Baseline (Day 1 of Week 0) to Week 96
Population: Intent to treat population: Participants who received at least 1 dose of study medication.Efavirenz group, 1 participant was excluded due to missing baseline CD4+ cell count.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Groups:
- TMC278 25mg: TMC278 25 mg once daily
Arm/Group | TMC278 25mg | TMC278 75 mg | TMC278 150 mg | All TMC278 | Efavirenz
Number analyzed (Participants) | 93 | 95 | 91 | 279 | 88
Cells per microliter | 145.9 (117.0) | 172.0 (156.5) | 158.9 (156.5) | 159.0 (144.4) | 159.8 (125.7)

8. Secondary Outcome: Change From Baseline in CD4+ Cell Count (Relative) at Week 96
Description: as for outcome 7
Time Frame: Baseline (Day 1 of Week 0) to Week 96
Population: Intent to treat (ITT) population: Participants who received at least 1 dose of study medication. Efavirenz group, 1 participant was excluded due to missing baseline CD4+ cell count.
Measure: Mean (Standard Deviation); unit: Percentage of CD4+ Cells
Arm/Group | TMC278 25mg | TMC278 75 mg | TMC278 150 mg | All TMC278 | Efavirenz
Number analyzed (Participants) | 93 | 95 | 91 | 279 | 88
Percentage of CD4+ Cells | 8.6 (6.9) | 9.9 (7.3) | 9.3 (7.1) | 9.3 (7.1) | 9.6 (7.0)

9. Secondary Outcome: Change From Baseline in CD4+ Cell Count (Absolute) at Week 240
Description: as for outcome 7
Time Frame: Baseline (Day 1 of Week 0) to Week 240
Population: ITT population: Participants who received at least 1 dose of study medication. Efavirenz group, 1 participant was excluded due to missing baseline CD4+ cell count. This was measured at Week 240 for the combined TMC278 and Efavirenz groups, as all TMC278 participants were switched after Week 96 initially to 75 mg and subsequently to 25 mg dose.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | All TMC278 | Efavirenz
Number analyzed (Participants) | 279 | 88
Cells per microliter | 221.0 (227.2) | 217.9 (213.7)

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count (Relative) at Week 240
Description: as for outcome 7
Time Frame: Baseline (Day 1 of week 0) to Week 240
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of CD4+ cells
Arm/Group | All TMC278 | Efavirenz
Number analyzed (Participants) | 279 | 88
Percentage of CD4+ cells | 8.7 (8.7) | 9.7 (9.1)

11. Secondary Outcome: Number of Participants With Virologic Failure for the Resistance Determinations by Developing Mutations: First Available On-Treatment Genotypic Data After Failure
Description: Virologic failure for the resistance determinations was defined as a viral load greater than 0.5 log10 copies /mL above the nadir with a minimum of 500 copies/mL. For this study, treatment-emergent mutations (for at least one treatment) are presented as Resistance associated mutation (RAMs): i) Non-nucleotide reverse transcriptase inhibitor (NNRTI) RAMs, ii) Nucleoside/tide reverse transcriptase inhibitor (N[t]RTI RAMs).
Time Frame: Week 240
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | All TMC278 | Efavirenz
Number analyzed (Participants) | 279 | 89
Participants
  Treatment-emergent NNRTI RAM | 17 | 4
  E138K | 7 | 0
  K101E | 6 | 0
  K103N | 1 | 3
  Treatment-emergent N(t)RTI RAM | 13 | 0
  M184V | 10 | 0

12. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hours (AUC24h) for TMC278
Description: For each participant, a single value for area under the plasma concentration-time curve from time of administration up to 24 hours post dosing (AUC24h) of TMC278 was estimated from a population pharmacokinetic model, based on all samples collected throughout the trial up to Week 96.
Time Frame: Up to Week 96
Population: Analysis included participants with sufficient number of pharmacokinetic samples in order to derive population pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TMC278 25 mg | TMC278 75 mg | TMC278 150 mg
Number analyzed (Participants) | 89 | 93 | 87
ng*h/mL | 2767 (1166) | 5906 (2419) | 10281 (4208)

13. Secondary Outcome: Trough Plasma Concentration (Ctrough) for TMC278
Description: For each participant, a single value for trough (i.e. predose) plasma concentration (Ctrough) of TMC278 was estimated from a population pharmacokinetic model, based on samples collected throughout the trial up to Week 96.
Time Frame: Up to Week 96
Population: Analysis included participants with sufficient number of pharnacokintetic samples in order to derive population pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC278 25 mg | TMC278 75 mg | TMC278 150 mg
Number analyzed (Participants) | 89 | 93 | 87
ng/mL | 92.7 (45.2) | 196.0 (90.1) | 342.0 (154.0)

14. Secondary Outcome: Number of Participants With Virologic Response (Viral Load Less Than 50 Copies Per mL) - as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm, by Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hours (AUC24h) Quartiles
Description: Quartile 1, 2, 3 and 4 of AUC24h means the quartile with the lowest 25%, 26-50%, 51-75% and the highest 25% of AUC24h values, respectively, irrespective of the different doses of TMC278. For each participant, a single value for area under the plasma concentration-time curve from time of administration up to 24 hours post dosing (AUC24h) of TMC278 was estimated from a population pharmacokinetic model, based on all samples collected throughout the trial up to Week 96. Virologic response was calculated by time to loss of virologic response (TLOVR) algorithm.
Time Frame: Up to Week 96
Population: Analysis included participants who received TMC278 with sufficient number of pharnacokintetic samples in order to derive population pharmacokinetic parameter. Participants who discontinued treatment for reasons other than virological failure were excluded from this analysis.
Measure: Number; unit: Participants
Groups:
- AUC24h Quartile 1; AUC24h Quartile 2; AUC24h Quartile 3; AUC24h Quartile 4: TMC278 25 mg, 75 mg, and 150 mg once daily
Arm/Group | AUC24h Quartile 1 | AUC24h Quartile 2 | AUC24h Quartile 3 | AUC24h Quartile 4
Number analyzed (Participants) | 58 | 54 | 59 | 56
Participants | 48 | 50 | 55 | 51

ADVERSE EVENTS:
Time Frame: Up to 336 weeks for participants in the TMC278 treatment group and up to 260 weeks for participants in the efavirenz treatment group.
Description: Adverse events were reported at Week 240 for the combined TMC278 and Efavirenz groups, as all TMC278 participants were switched after Week 96 initially to 75 mg and subsequently to 25 mg dose.
Arm/Group | All TMC278 | Efavirenz
Serious Adverse Events (participants affected / at risk) | 49/279 | 17/89
Other Adverse Events (participants affected / at risk) | 241/279 | 82/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All TMC278 (N=279) | Efavirenz (N=89)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Meningitis tuberculous (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Perianal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood amylase increased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Chondrosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Ovarian cystectomy (Surgical and medical procedures) | 1 | 0
Penile prosthesis insertion (Surgical and medical procedures) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All TMC278 (N=279) | Efavirenz (N=89)
Anaemia (Blood and lymphatic system disorders) | 24 | 2
Vertigo (Ear and labyrinth disorders) | 4 | 10
Conjunctivitis (Eye disorders) | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 20 | 4
Abdominal pain upper (Gastrointestinal disorders) | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 33 | 16
Dyspepsia (Gastrointestinal disorders) | 36 | 7
Haemorrhoids (Gastrointestinal disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 100 | 26
Vomiting (Gastrointestinal disorders) | 33 | 11
Fatigue (General disorders) | 23 | 4
Pyrexia (General disorders) | 19 | 3
Body tinea (Infections and infestations) | 4 | 7
Bronchitis (Infections and infestations) | 20 | 3
Condyloma acuminatum (Infections and infestations) | 17 | 3
Gastroenteritis (Infections and infestations) | 11 | 5
Herpes simplex (Infections and infestations) | 25 | 7
Herpes zoster (Infections and infestations) | 15 | 4
Influenza (Infections and infestations) | 27 | 8
Nasopharyngitis (Infections and infestations) | 45 | 19
Pharyngitis (Infections and infestations) | 18 | 4
Respiratory tract infection (Infections and infestations) | 9 | 5
Respiratory tract infection viral (Infections and infestations) | 1 | 7
Rhinitis (Infections and infestations) | 12 | 5
Sinusitis (Infections and infestations) | 20 | 3
Tinea pedis (Infections and infestations) | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 49 | 9
Urinary tract infection (Infections and infestations) | 21 | 6
Alanine aminotransferase increased (Investigations) | 21 | 6
Aspartate aminotransferase increased (Investigations) | 17 | 5
Blood cholesterol increased (Investigations) | 13 | 11
Low density lipoprotein increased (Investigations) | 16 | 9
Anorexia (Metabolism and nutrition disorders) | 19 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 3
Dizziness (Nervous system disorders) | 31 | 27
Headache (Nervous system disorders) | 62 | 15
Somnolence (Nervous system disorders) | 10 | 10
Abnormal dreams (Psychiatric disorders) | 6 | 5
Depression (Psychiatric disorders) | 19 | 9
Insomnia (Psychiatric disorders) | 23 | 6
Nightmare (Psychiatric disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 7
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 7 | 5
Hypertension (Vascular disorders) | 22 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days